CLINICAL TRIAL: NCT02265458
Title: Musical Intervention in the ICU: Effect on Tolerance and Acceptance of Non-invasive Ventilation
Brief Title: Musical Intervention in Non-invasive Ventilation
Acronym: Mus-IRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P131201
Record Dates: First submitted 2014-08-25; First posted 2014-10-16 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Respiratory Failure
Keywords: Respiratory failure; NIV; Musical intervention
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Musical intervention and sensory isolation (Experimental): 30 minutes musical intervention during NIV will be administrated, along with sensory isolation (mask obscuring the eyes)
  Interventions: Behavioral: Musical intervention and sensory isolation
- Sensory isolation (Active Comparator): Sensory isolation
  Interventions: Behavioral: Musical intervention and sensory isolation
- Standard of care (No Intervention): Standard of care

INTERVENTIONS:
Behavioral: Musical intervention and sensory isolation — 30 minutes musical intervention during NIV will be administrated, along with sensory isolation (mask obscuring the eyes)
  Arms: Musical intervention and sensory isolation; Sensory isolation

SUMMARY:
Non-invasive ventilation (NIV) might be associated with anxiety, thus leading to NIV failure, and intubation. Music therapy has been used in various clinical context, including in ICU patients under mechanical ventilation. We aim to evaluate the effect of a musical intervention on respiratory comfort during NIV for acute respiratory failure.

DETAILED DESCRIPTION:
We plan a randomized controlled trial with 3 different arms, in ICU patients requiring NIV for acute respiratory failure : "usual care", "sensory isolation" and "sensory isolation and musical intervention".At the onset of respiratory failure, each patient will be randomized in one of the 3 arms. "Usual care" assigned patients will receive NIV according to each unit protocol; "sensory isolation" assigned patients will receive NIV associated with a mask obscuring the eyes and a noise-reducing headset."musical intervention patients" will receive a 30 minutes musical intervention during each NIV session. Respiratory discomfort will be blindly assessed before, immediately after NIV is correctly set (5 minutes), at 30 minutes, and at hours 1, 2, 3, 4, 6, 8, 12, 16, 20, 24 according to NIV session length, and at the end of NIV session during each NIV session.

ELIGIBILITY:
Inclusion Criteria:

* respiratory distress requiring NIV
* Glasgow coma score above 12

Exclusion Criteria:

* NIV contraindication : Hemodynamic failure, neurologic failure, head trauma, vomiting
* Severe hypoacusis people without hearing device
* Decision to limit active treatment with an estimated life expectancy of less than 48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2015-05; Primary Completion 2016-10 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Variation of respiratory discomfort during the 30 first minutes of NIV | 30 minutes
  Measure of respiratory discomfort at the beginning and the end of the first NIV session, with an analogic visual scale.

SECONDARY OUTCOMES:
Evolution of respiratory parameters | participants will be followed for the duration of hospital stay or maximum 28 days
  Measure of respiratory rate
Evolution of respiratory parameters | participants will be followed for the duration of hospital stay or maximum 28 days
  Transcutaneous oxygen saturation
Evolution of respiratory parameters | participants will be followed for the duration of hospital stay or maximum 28 days
  Respiratory tidal volume
Number of NIV failure | participants will be followed for the duration of hospital stay or maximum 28 days
  NIV failure
Quality of life | 3 months
  Questionnaire
Evolution of cardiovascular parameters | participants will be followed for the duration of hospital stay or maximum 28 days
  Measure of heart rate
Evolution of cardiovascular parameters | participants will be followed for the duration of hospital stay or maximum 28 days
  Measure of blood pressure
Post traumatic stress disorder | 3 months
  questionnaire
overall assessment of NIV (in terms of discomfort, satisfaction, and trauma) | 3 months
  Questionnaire (scale)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan MESSIKA, MD, Principal Investigator — AP-HP Louis Mourier
Locations (3):
- France (3):
  - Hôpital Louis Mourier, Colombes
  - CHD Vendée, La Roche-sur-Yon
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Messika J, Hajage D, Panneckoucke N, Villard S, Martin Y, Renard E, Blivet A, Reignier J, Maquigneau N, Stoclin A, Puechberty C, Guetin S, Dechanet A, Fauquembergue A, Gaudry S, Dreyfuss D, Ricard JD. Effect of a musical intervention on tolerance and efficacy of non-invasive ventilation in the ICU: study protocol for a randomized controlled trial (MUSique pour l'Insuffisance Respiratoire Aigue - Mus-IRA). Trials. 2016 Sep 13;17(1):450. doi: 10.1186/s13063-016-1574-z. PMID 27618935